CLINICAL TRIAL: NCT05917860
Title: Effect of Neoadjuvant Degarelix on MRI-guided Transurethral Ultrasound Ablation (TULSA) in Patients with Intermediate-risk Prostate Cancer: a Pilot Study
Brief Title: Neoadjuvant ADT with TULSA in the Treatment of Intermediate Risk Prostate Cancer
Acronym: NeoADT-TULSA
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T1338/2023
Record Dates: First submitted 2023-05-02; First posted 2023-06-26 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Localized Prostate Carcinoma; Castration-Naive Prostate Cancer; Intermediate Risk Prostate Cancer; Prostate Cancer
Keywords: MRI-guided transurethral ultrasound ablation; Androgen deprivation therapy; Neoadjuvant androgen deprivation therapy; TULSA; Prostate cancer; Thermal ablation; Therapeutic ultrasound; Ablation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Intervention Model Description: Procedure: Magnetic resonance imaging-guided transurethral ultrasound ablation of the prostate (TULSA)
  Drug: Degarelix
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 3-month neoadjuvant Degarelix followed by whole-gland MRI-guided transurethral ultrasound ablation (Experimental): After three months of neoadjuvant ADT with Degarelix, the subject will undergo whole-prostate gland MRI-guided transurethral ultrasound ablation (TULSA) (TULSA-PRO, Profound Medical Inc., Toronto, Canada) treatment.
  Interventions: Drug: Degarelix; Device: MRI-guided transurethral ultrasound ablation (TULSA)

INTERVENTIONS:
Drug: Degarelix — Degarelix is injected subcutaneously into the fatty tissue of the abdomen. A typical protocol consists of a starting dose of 240 mg with a maintenance dose of 80 mg administered every 28 days. In this study, one starting dose and two maintenance doses of Degarelix will be administered between baseline and TULSA treatment in accordance with the terms of Degarelix marketing authorizations.
  Other Names: Firmagon
Device: MRI-guided transurethral ultrasound ablation (TULSA) — MRI-guided transurethral ultrasound ablation (TULSA) (TULSA-PRO, Profound Medical Inc., Toronto, Canada) will be used to deliver whole-prostate gland treatment in accordance with the terms of TULSA marketing authorizations. The treating physicians will contour the entire prostate gland for a whole gland ablation.
  Other Names: TULSA-PRO

SUMMARY:
Clinical studies have shown that magnetic resonance imaging-guided transurethral ultrasound ablation (TULSA) of the prostate is safe and effective. In the TULSA procedure, prostate tissue is killed by heating with ultrasound. This clinical trial explores if adding drug therapy with Degarelix before TULSA has the potential to improve further the effectiveness of TULSA in the treatment of localized prostate cancer, especially for patients with more aggressive diseases.

DETAILED DESCRIPTION:
Androgen deprivation therapy (ADT) has been shown to reduce prostate and tumor size. In this study, magnetic resonance imaging (MRI) is used to investigate the effect of Degarelix ADT on the properties of prostate tissue that can affect the heating of the tissues in the TULSA procedure. The main goal is to find out if ADT can change the tissue structure in a way that improves the ability of the TULSA procedure to heat tissues and better kill the diseased tissue, reducing the chance of the disease reoccurring. ADT and the TULSA procedure can help patients with more aggressive diseases avoid the adverse effects associated with surgery or radiation therapy. Specific objectives are:

1. To measure the change in prostate and tumor size, tissue structural changes, and the blood flow within the prostate after ADT.
2. To measure the distribution of heating over the prostate after TULSA treatment.
3. To evaluate complications and genitourinary function and quality of life with patient-reported outcome measures.
4. To evaluate local cancer control and longer-term oncological outcomes after combination therapy of neoadjuvant ADT and TULSA treatment.

About 15 subjects will participate. Each will receive Degarelix for three months, followed by whole-prostate gland TULSA treatment, and be followed for five years. Throughout the study, subjects will receive MRI scans and complete questionnaires regarding functional status and quality of life to understand the side effects.

ELIGIBILITY:
Inclusion Criteria:

* Male age ≥ 40 years and candidate for radical prostate cancer treatment
* Estimated life expectancy > 8 years
* At least one MRI-visible and biopsy-concordant tumor defined as Prostate Imaging-Reporting and Data System v2 (PI-RADS v2.1) ≥ 3
* Biopsy-confirmed, intermediate-risk localized prostate cancer:
* Clinical or radiological tumor stage ≤ T2c, N0, M0
* ISUP GG 2 or 3
* Biopsy obtained ≥ 6 weeks and ≤ 12 months before treatment
* PSA ≤ 20 ng/ml
* No prior definitive treatment of prostate cancer
* Eligible for MRI
* Eligible for general anesthesia (American Society of Anesthesiologists Class III or less)
* Patients taking 5-alpha reductase inhibitors (5-ARIs) are eligible if use is discontinued three months before and throughout the study period.
* Informed consent: The patient must speak Finnish, English, or Swedish and must be able to understand the meaning of the study. The patient must be willing and able to sign the appropriate Ethics Committee (EC) approved informed consent documents in the presence of the designated staff.

Exclusion Criteria:

* Prior prostate cancer treatment with chemotherapy or hormonal therapy, including chemical or surgical castration, antiandrogen therapy, or androgen-receptor signaling inhibitors.
* Relative or absolute contraindication to Degarelix
* Severe, active cardiovascular comorbidity including unstable angina pectoris, congestive heart failure, deep vein thrombosis, pulmonary embolism, or myocardial infarction within the last six months.
* Inability to undergo MRI due to claustrophobia or contraindications (cardiac pacemaker, intracranial clips, etc.)
* Severe kidney failure as determined by estimated glomerular filtration rate (eGFR) less than 30 ml/min per 1.73 m2
* Prostate calcifications obstructing the planned ultrasound beam path in the line of sight of the MRI visible tumor
* Prostate cysts at the prostate capsule within the planned ultrasound beam path in the line of sight of the MRI visible tumor
* Evidence of extraprostatic disease based on imaging (MRI, bone scintigraphy, single-photon emission tomography, computed tomography, prostate-specific membrane antigen-positron emission tomography [PSMA-PET]) or histopathology
* History of chronic inflammatory conditions (e.g., inflammatory bowel disease) affecting the rectum (also includes rectal fistula and anal/rectal stenosis)
* Hip replacement surgery or other metal in the pelvic area
* Known allergy or contraindication to gadolinium or gastro-intestinal anti-spasmodic drug glucagon
* Concomitant treatment with medications contraindicated to Glucagen used as antispasmolytic agent during TULSA treatment (e.g., Feochromocytoma)
* Any other conditions that might compromise patient safety, based on the clinical judgment of the responsible urologist
* Another primary malignancy unless disease-free survival is > 8 years

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in prostate volume after neoadjuvant ADT | Baseline and four, eight, and 12 weeks of ADT.
  The prostate volume change will be determined by comparing the prostate volume measured on T2-weighted MRI at four, eight, and 12 weeks of ADT to that at baseline.
Change in prostate tumor volume after neoadjuvant ADT | Baseline and four, eight, and 12 weeks of ADT.
  The prostate tumor volume change will be determined by comparing the prostate tumor volume measured on T2-weighted MRI at four, eight, and 12 weeks of ADT to that at baseline.
The frequency and severity of adverse events | Every follow-up visit until the first year of follow-up.
  The frequency and severity of adverse events after neoadjuvant Degarelix and TULSA treatment will be determined by using the CTCAE v6.0 classification. Adverse events attributed to TULSA will also be graded using the Clavien Dindo classification for surgical complications.

SECONDARY OUTCOMES:
Change in prostate tumor-capsule contact length after neoadjuvant ADT | Baseline and four, eight, and 12 weeks of ADT.
  The prostate tumor-capsule contact length change will be determined by comparing the prostate tumor-capsule contact length measured on T2-weighted MRI at four, eight, and 12 weeks of ADT to that at baseline.
Change in prostate vascular perfusion after neoadjuvant ADT | Baseline and four, eight, and 12 weeks of ADT.
  The change in prostate vascular perfusion will be determined by comparing average blood flow values in the prostate measured on dynamic contrast-enhanced T1-weighted MRI at four, eight, and 12 weeks of ADT to that at baseline.
Change in prostate tumor vascular perfusion after neoadjuvant ADT | Baseline and four, eight, and 12 weeks of ADT.
  The change in prostate tumor vascular perfusion will be determined by comparing average blood flow values in the prostate tumor measured on dynamic contrast-enhanced T1-weighted MRI at four, eight, and 12 weeks of ADT to that at baseline.
Change in periprostatic, prostate and tumor tissue structures after neoadjuvant ADT | Baseline and four, eight, and 12 weeks of ADT.
  The change in periprostatic, prostate and tumor tissue structures will be determined by comparing the radiomics features extracted from T2-weighted, T2 relaxation time mapping, and diffusion-weighted images at four, eight, and 12 weeks of ADT to that at baseline.
Thermal coverage after whole-prostate gland TULSA | Immediately after the TULSA procedure.
  Thermal coverage of the target volume achieved by whole-prostate gland TULSA will be determined by comparing physician-defined target boundaries to MRI measurements of temperature distributions, thermal dose distributions, and acute treatment-induced perfusion defect immediately post-treatment.
Change in quality of life (QoL) and functional status outcomes after neoadjuvant ADT | Baseline and 12 weeks of ADT.
  The change in QoL and functional status outcomes will be determined by comparing the summary scores of urinary incontinence, urinary irritative/obstructive, bowel, sexual and hormonal domains of the Expanded Prostate Index Composite-26 (EPIC-26) questionnaire at 12 weeks of ADT to that at baseline. EPIC-26 contains 26 items with response options for each EPIC item forming a Likert Scale, and multi-item scale scores transformed linearly to a 0-100 scale, with higher scores representing better functional status/QoL.
Change in lower urinary tract symptoms after neoadjuvant ADT | Baseline and 12 weeks of ADT.
  The change in lower urinary tract symptoms will be determined by comparing the International Prostate Symptom Score (IPSS) at 12 weeks of ADT to that at baseline. The possible scores for the IPSS questionnaire range from 0 to 35, with higher scores representing worse symptoms.
Change in erectile function after neoadjuvant ADT | Baseline and 12 weeks of ADT.
  The change in erectile function will be determined by comparing the International Index of Erectile Function (IIEF-5) score at 12 weeks of ADT to that at baseline. The possible scores for the IIEF-5 range from 5 to 25, with higher scores representing a better erectile function.
Change in quality of life (QoL) and functional status outcomes after neoadjuvant ADT and whole-prostate gland TULSA | Baseline and 12 weeks of ADT, and three, six, 12, 36 and 60 months after the TULSA procedure.
  The change in QoL and functional status outcomes will be determined by comparing the summary scores of urinary incontinence, urinary irritative/obstructive, bowel, sexual and hormonal domains of the Expanded Prostate Index Composite (EPIC-26) questionnaire at three, six, 12, 36 and 60 months post-TULSA to that at baseline and TULSA procedure. EPIC-26 contains 26 items with response options for each EPIC item forming a Likert Scale, and multi-item scale scores transformed linearly to a 0-100 scale, with higher scores representing better functional status/QoL.
Change in lower urinary tract symptoms after neoadjuvant ADT and whole-prostate gland TULSA | Baseline and 12 weeks of ADT, and three, six, 12, 36 and 60 months after the TULSA procedure.
  The change in lower urinary tract symptoms will be determined by comparing the International Prostate Symptom Score (IPSS) at three, six, 12, 36 and 60 months post-TULSA to that at baseline and TULSA procedure. The possible scores for the IPSS questionnaire range from 0 to 35, with higher scores representing worse symptoms.
Change in erectile function after neoadjuvant ADT and whole-prostate gland TULSA | Baseline and 12 weeks of ADT, and three, six, 12, 36 and 60 months after the TULSA procedure.
  The change in erectile function will be determined by comparing the International Index of Erectile Function (IIEF-5) score at three, six, 12, 36 and 60 months post-TULSA to that at baseline and TULSA procedure. The possible scores for the IIEF-5 range from 5 to 25, with higher scores representing a better erectile function.
The frequency and severity of adverse events during extended follow-up | Every follow-up visit until the five years of follow-up.
  The frequency and severity of adverse events after neoadjuvant Degarelix and TULSA treatment will be determined using the CTCAE v6.0 classification. Adverse events attributed to TULSA will also be graded using the Clavien Dindo classification for surgical complications.
Salvage therapy-free survival | Every post-TULSA follow-up visit until the five years of follow-up.
  Salvage therapy-free survival will be defined as freedom from radical salvage treatments for prostate cancer including radical prostatectomy, radiotherapy, or ablation, and reported as the proportion of subjects who have not reached those events.
Systemic therapy-free survival | Every post-TULSA follow-up visit until the five years of follow-up.
  Systemic therapy-free survival will be defined as freedom from additional systemic therapy including but not limited to additional ADT or chemotherapy for the treatment of prostate cancer, and reported as the proportion of subjects who have not reached those events.
Failure-free survival | Every post-TULSA follow-up visit until the five years of follow-up.
  Failure-free survival will be defined as freedom from salvage treatment, systemic treatment, metastases, or death from prostate cancer, and reported as the proportion of subjects who have not reached those events.
Metastasis-free, prostate cancer-specific, and overall survival | One, three and five years after the TULSA procedure.
  Metastasis-free, prostate cancer-specific and overall survivals will be assessed one, three, and five years after TULSA and reported as the proportion of subjects who have not reached those endpoints.
Biochemical failure-free survival | One, three, and five years after the TULSA procedure.
  PSA at each timepoint, as well as PSA nadir, will be reported. The proportion of subjects with biochemical failure, defined as a PSA value more than 2.0 ng/ml above nadir, will be reported.
Freedom from biopsy-proven clinically-significant prostate cancer | Twelve months after the TULSA procedure
  Histopathologic verification of treatment response to TULSA treatment will be confirmed at 12 months post-TULSA with targeted plus 10-12-core systematic biopsy. The proportion of subjects with a clinically-significant disease, defined as Gleason grade ≥ 3 + 4 and ISUP (International Society of Urological Pathology) grade group ≥ 2 prostate cancer, on biopsy, will be reported.
Freedom from any biopsy-proven prostate cancer | Twelve months after the TULSA procedure
  Histopathologic verification of treatment response to TULSA treatment will be confirmed at 12 months post-TULSA with targeted plus 10-12-core systematic biopsy. The number, location, grade, and percent of cancer involvement within each core will be collected. The proportion of subjects with any prostate cancer on biopsy, will be reported.

OTHER OUTCOMES:
Change in prostate volume after whole-prostate gland TULSA | Three and twelve months after TULSA procedure
  The prostate volume change will be determined by comparing the prostate volume measured on T2-weighted MRI at three, and 12 months after TULSA to that at TULSA procedure.
Change in maximum urinary flow rate after neoadjuvant ADT and whole-gland TULSA | Baseline, 12 weeks of ADT, and three, 12, 36 and 60 months after the TULSA procedure
  The change in maximum urinary flow rate (Qmax) (ml/s) will be determined by comparing Qmax values at 12 weeks of ADT and three, 12, 36, and 60 months post-TULSA to that at baseline and TULSA procedure.
Change in average urinary flow rate after neoadjuvant ADT and whole-gland TULSA | Baseline, 12 weeks of ADT, and three, 12, 36 and 60 months after the TULSA procedure
  The change in average urinary flow rate (ml/s) will be determined by comparing average flow rate values at 12 weeks of ADT and three, 12, 36, and 60 months post-TULSA to that at baseline and TULSA procedure.
Change in post-void residual volume after neoadjuvant ADT and whole-gland TULSA | Baseline, 12 weeks of ADT, and three, 12, 36 and 60 months after the TULSA procedure
  The change in post-void residual volume (PVR) (ml) will be determined by comparing PVR values at 12 weeks of ADT and three, 12, 36, and 60 months post-TULSA to that at baseline and TULSA procedure.
Change in voided volume after neoadjuvant ADT and whole-gland TULSA | Baseline, 12 weeks of ADT, and three, 12, 36 and 60 months after the TULSA procedure
  The change in voided volume (ml) will be determined by comparing voided volume values at 12 weeks of ADT and three, 12, 36, and 60 months post-TULSA to that at baseline and TULSA procedure.
Freedom from any suspicious lesion on MRI | Three and twelve months after the TULSA procedure
  3T prostate multiparametric MRI three and twelve months after TULSA treatment will be assessed for residual or recurrent disease according to the Prostate Imaging for Recurrence Reporting (PI-RR) system guidelines. The proportion of subjects with a suspicious lesion on MRI, defined as lesion ≥ PI-RR 3, will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael HJ Anttinen, MD, PhD, Principal Investigator — Department of Urology, University of Turku and Turku University Hospital, Turku, Finland
Locations (1):
- Turku University Hospital, Turku, Southwest Finland, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anttinen M, Blanco Sequeiros R, Bostrom PJ, Taimen P. Evolving imaging methods of prostate cancer and the emergence of magnetic resonance imaging guided ablation techniques. Front Oncol. 2022 Nov 17;12:1043688. doi: 10.3389/fonc.2022.1043688. eCollection 2022. PMID 36465377
- [Background] Valerio M, Cerantola Y, Eggener SE, Lepor H, Polascik TJ, Villers A, Emberton M. New and Established Technology in Focal Ablation of the Prostate: A Systematic Review. Eur Urol. 2017 Jan;71(1):17-34. doi: 10.1016/j.eururo.2016.08.044. Epub 2016 Aug 29. PMID 27595377
- [Background] Klotz L, Pavlovich CP, Chin J, Hatiboglu G, Koch M, Penson D, Raman S, Oto A, Futterer J, Serrallach M, Relle J, Lotan Y, Heidenreich A, Bonekamp D, Haider M, Tirkes T, Arora S, Macura KJ, Costa DN, Persigehl T, Pantuck AJ, Bomers J, Burtnyk M, Staruch R, Eggener S. Magnetic Resonance Imaging-Guided Transurethral Ultrasound Ablation of Prostate Cancer. J Urol. 2021 Mar;205(3):769-779. doi: 10.1097/JU.0000000000001362. Epub 2020 Oct 6. PMID 33021440
- [Background] EAU Guidelines 2023, presented at the EAU Annual Congress Milan 2023. ISBN 978-94-92671-16-5.
- [Background] Denham JW, Steigler A, Lamb DS, Joseph D, Turner S, Matthews J, Atkinson C, North J, Christie D, Spry NA, Tai KH, Wynne C, D'Este C. Short-term neoadjuvant androgen deprivation and radiotherapy for locally advanced prostate cancer: 10-year data from the TROG 96.01 randomised trial. Lancet Oncol. 2011 May;12(5):451-9. doi: 10.1016/S1470-2045(11)70063-8. PMID 21440505
- [Background] Hu J, Xu H, Zhu W, Wu F, Wang J, Ding Q, Jiang H. Neo-adjuvant hormone therapy for non-metastatic prostate cancer: a systematic review and meta-analysis of 5,194 patients. World J Surg Oncol. 2015 Feb 22;13:73. doi: 10.1186/s12957-015-0503-z. PMID 25884478
- [Background] Nishiyama T. Serum testosterone levels after medical or surgical androgen deprivation: a comprehensive review of the literature. Urol Oncol. 2014 Jan;32(1):38.e17-28. doi: 10.1016/j.urolonc.2013.03.007. Epub 2013 Jun 13. PMID 23769268
- [Background] Christie DRH, Mitina N, Sharpley CF. A prospective study of the effect of testosterone escape on preradiotherapy prostate-specific antigen kinetics in prostate cancer patients undergoing neoadjuvant androgen deprivation therapy. Curr Urol. 2021 Mar;15(1):63-67. doi: 10.1097/CU9.0000000000000008. Epub 2021 Mar 29. PMID 34084124
- [Background] Klotz LH, Goldenberg SL, Jewett MA, Fradet Y, Nam R, Barkin J, Chin J, Chatterjee S; Canadian Uro-Oncology Group. Long-term followup of a randomized trial of 0 versus 3 months of neoadjuvant androgen ablation before radical prostatectomy. J Urol. 2003 Sep;170(3):791-4. doi: 10.1097/01.ju.0000081404.98273.fd. PMID 12913699
- [Background] Kumar S, Shelley M, Harrison C, Coles B, Wilt TJ, Mason MD. Neo-adjuvant and adjuvant hormone therapy for localised and locally advanced prostate cancer. Cochrane Database Syst Rev. 2006 Oct 18;2006(4):CD006019. doi: 10.1002/14651858.CD006019.pub2. PMID 17054269
- [Background] Sumitomo M, Hayashi M, Watanabe T, Tsugawa M, Noma H, Yamaguchi A, Nagakura K, Hayakawa M, Uchida T. Efficacy of short-term androgen deprivation with high-intensity focused ultrasound in the treatment of prostate cancer in Japan. Urology. 2008 Dec;72(6):1335-40. doi: 10.1016/j.urology.2007.12.041. Epub 2008 Mar 20. PMID 18355899
- [Background] Aoyagi, Teiichiro, and Isao Kuroda. Enhancement of HIFU Effect by Simultaneous Short Course Degarelix for Early Stage Prostate Cancer: A Pilot Study. Open Journal of Urology 6.03 (2016): 49-54.
- [Background] Crawford ED, Shore ND, Moul JW, Tombal B, Schroder FH, Miller K, Boccon-Gibod L, Malmberg A, Olesen TK, Persson BE, Klotz L. Long-term tolerability and efficacy of degarelix: 5-year results from a phase III extension trial with a 1-arm crossover from leuprolide to degarelix. Urology. 2014 May;83(5):1122-8. doi: 10.1016/j.urology.2014.01.013. Epub 2014 Mar 22. PMID 24661333
- [Background] Anttinen M, Makela P, Viitala A, Nurminen P, Suomi V, Sainio T, Saunavaara J, Taimen P, Sequeiros RB, Bostrom PJ. Salvage Magnetic Resonance Imaging-guided Transurethral Ultrasound Ablation for Localized Radiorecurrent Prostate Cancer: 12-Month Functional and Oncological Results. Eur Urol Open Sci. 2020 Nov 25;22:79-87. doi: 10.1016/j.euros.2020.10.007. eCollection 2020 Dec. PMID 34337481
- [Background] Anttinen M, Makela P, Nurminen P, Yli-Pietila E, Suomi V, Sainio T, Saunavaara J, Taimen P, Blanco Sequeiros R, Bostrom PJ. Palliative MRI-guided transurethral ultrasound ablation for symptomatic locally advanced prostate cancer. Scand J Urol. 2020 Dec;54(6):481-486. doi: 10.1080/21681805.2020.1814857. Epub 2020 Sep 8. PMID 32897169
- [Background] Dora C, Clarke GM, Frey G, Sella D. Magnetic Resonance Imaging-Guided Transurethral Ultrasound Ablation of Prostate Cancer: A Systematic Review. J Endourol. 2022 Jun;36(6):841-854. doi: 10.1089/end.2021.0866. Epub 2022 Mar 7. PMID 35029127
- [Background] Pooli A, Johnson DC, Shirk J, Markovic D, Sadun TY, Sisk AE Jr, Mohammadian Bajgiran A, Afshari Mirak S, Felker ER, Hughes AK, Raman SS, Reiter RE. Predicting Pathological Tumor Size in Prostate Cancer Based on Multiparametric Prostate Magnetic Resonance Imaging and Preoperative Findings. J Urol. 2021 Feb;205(2):444-451. doi: 10.1097/JU.0000000000001389. Epub 2020 Oct 7. PMID 33026934
- [Background] Bjoreland U, Nyholm T, Jonsson J, Skorpil M, Blomqvist L, Strandberg S, Riklund K, Beckman L, Thellenberg-Karlsson C. Impact of neoadjuvant androgen deprivation therapy on magnetic resonance imaging features in prostate cancer before radiotherapy. Phys Imaging Radiat Oncol. 2021 Feb 24;17:117-123. doi: 10.1016/j.phro.2021.01.004. eCollection 2021 Jan. PMID 33898790
- [Background] Washino S, Hirai M, Saito K, Kobayashi Y, Arai Y, Miyagawa T. Impact of Androgen Deprivation Therapy on Volume Reduction and Lower Urinary Tract Symptoms in Patients with Prostate Cancer. Low Urin Tract Symptoms. 2018 Jan;10(1):57-63. doi: 10.1111/luts.12142. Epub 2016 Dec 12. PMID 27943566
- [Background] Hotker AM, Mazaheri Y, Zheng J, Moskowitz CS, Berkowitz J, Lantos JE, Pei X, Zelefsky MJ, Hricak H, Akin O. Prostate Cancer: assessing the effects of androgen-deprivation therapy using quantitative diffusion-weighted and dynamic contrast-enhanced MRI. Eur Radiol. 2015 Sep;25(9):2665-72. doi: 10.1007/s00330-015-3688-1. Epub 2015 Mar 29. PMID 25820537
- [Background] Marra G, Dell'oglio P, Baghdadi M, Cathelineau X, Sanchez-Salas R; EvaluatioN of HIFU Hemiablation and short-term AndrogeN deprivation therapy Combination to Enhance prostate cancer control (ENHANCE) Study. Multimodal treatment in focal therapy for localized prostate cancer using concomitant short-term androgen deprivation therapy: the ENHANCE prospective pilot study. Minerva Urol Nefrol. 2019 Oct;71(5):544-548. doi: 10.23736/S0393-2249.19.03599-9. Epub 2019 Sep 6. PMID 31508924
- See also: Turku HIFU research centre — http://hifu.utu.fi